CLINICAL TRIAL: NCT07342712
Title: A Phase ⅢB Clinical Trial Evaluating the Long-term Effects of Gecacitinib Treatment on Myelofibrosis and Gene Mutation Levels in Patients Previously Enrolled in Clinical Trails of Gecacitinib for the Treatment of Myelofibrosis
Brief Title: Clinical Trail to Evaluate the Effect of Long-term Treatment With Gecacitinib on Myelofibrosis and Gene Mutation Levels
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20250082B-R2
Record Dates: First submitted 2025-07-04; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was an observational study, and about 40 patients with intermediate and high risk myelofibrosis who had participated in any previous clinical study of Gecacitinib hydrochloride and were still receiving Gecacitinib treatment in our center were expected to be enrolled. There was no additional drug intervention, only the myelofibrosis grade and gene mutation level of the patients were collected. Subjects who met all inclusion criteria and none of the exclusion criteria were eligible for inclusion in this study. After informed consent was obtained and screening was successful, bone marrow aspiration, bone marrow biopsy, and gene mutation testing were performed once. If bone marrow was extracted, peripheral blood could be used for gene mutation testing, and then annually until the permanent discontinuation of Gecacitinib.

DETAILED DESCRIPTION:
Previous clinical trials of Gecacitinib hydrochloride tablets in the treatment of myelofibrosis initiated by our center include: 1) ZGJAK002 trial (NCT03886415) : A multicenter phase Ⅱ clinical trial of the safety and efficacy of 100mg BID and 200mg QD of Gecacitinib in the treatment of intermediate and high risk myelofibrosis (n=118). 2) ZGJAK006 study (NCT04217993) : a phase ⅡB clinical trial of the safety and efficacy of gefitinib in Ruxolitinib intolerant myelofibrosis patients (n=51); 3) ZGJAK017 study (NCT04851535) : a phase Ⅱ trial (n=34) to evaluate the efficacy and safety of Gecacitinib in Ruxolitinib refractory or relapsed myelofibrosis patients; 4) ZGJAK016 trial (NCT04617028) : a randomized, double-blind, double-dummy, parallel-controlled, multicenter phase III trial (n=105). At present, the follow-up of the project has ended and the Gecacitinib donation phase has begun.

This study was an observational study, and about 40 patients with intermediate and high risk myelofibrosis who had participated in any previous clinical study of Gecacitinib hydrochloride and were still receiving Gecacitinib treatment in our center were expected to be enrolled. There was no additional drug intervention, only the myelofibrosis grade and gene mutation level of the patients were collected. Subjects who met all inclusion criteria and none of the exclusion criteria were eligible for inclusion in this study. After informed consent was obtained and screening was successful, bone marrow aspiration, bone marrow biopsy, and gene mutation testing were performed once. If bone marrow was extracted, peripheral blood could be used for gene mutation testing, and then annually until the permanent discontinuation of Gecacitinib.

The primary objective was to evaluate the myelofibrosis grade in patients with MF who had previously participated in a clinical study of Gecacitinib and were still receiving gefitinib. The secondary objective was to evaluate the change from baseline in JAK2 isomutations.

ELIGIBILITY:
Inclusion Criteria:

* They had been enrolled in previous clinical trials of gefitinib for myelofibrosis (ZGJAK002, ZGJAK006, ZGJAK016 and ZGJAK017) and were still receiving gefitinib treatment.
* Comply with the requirements of the ethics committee, voluntarily sign the informed consent.
* Able to adhere to study and follow-up procedures.

Exclusion Criteria:

* Patients with other serious diseases that the researcher believes may affect patient compliance and outcome observation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was an observational study, and about 40 patients with intermediate and high risk myelofibrosis who had participated in any previous clinical study of Gecacitinib hydrochloride and were still receiving Gecacitinib treatment in our center were expected to be enrolled. There was no additional drug intervention, only the myelofibrosis grade and gene mutation level of the patients were collected. Subjects who met all inclusion criteria and none of the exclusion criteria were eligible for inclusion in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-12-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with worsening/stable/improving myelofibrosis grade after treatment | Successfully enrolled patients will undergo bone marrow biopsy as indicated by follow-up, and then once per 1 year until Gecacitinib is permanently discontinued or assessed up to 5 years, whichever came first.
  Sample collection: Bone marrow biopsy tissue was at least 1.5 cm in length to ensure accuracy of bone marrow analysis. The bone marrow fibers were graded by silver staining to ensure the objectivity and reproducibility of the grading results

SECONDARY OUTCOMES:
The changes of JAK2 V617F, CALR and MPL W515L/K gene mutations after treatment were compared with those before treatment | Successfully enrolled patients will undergo genetic testing as indicated by follow-up, and then once per 1 year until Gecacitinib is permanently discontinued or assessed up to 5 years, whichever came first.
  Sample collection: Approximately 3-5 mL of forearm venous blood was collected to ensure adequate blood volume for molecular biological quantitative analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zhang Y, Zhou H, Jiang Z, Wu D, Zhuang J, Li W, Jiang Q, Wang X, Huang J, Zhu H, Yang L, Du X, Li F, Xia R, Zhang F, Hu J, Li Y, Hu Y, Liu J, Jin C, Sun K, Zhou Z, Wu L, Yu W, Jin J. Safety and efficacy of jaktinib in the treatment of Janus kinase inhibitor-naive patients with myelofibrosis: Results of a phase II trial. Am J Hematol. 2022 Dec;97(12):1510-1519. doi: 10.1002/ajh.26709. Epub 2022 Oct 4. PMID 36054786
- [Background] Zhang Y, Zhou H, Duan M, Gao S, He G, Jing H, Li J, Ma L, Zhu H, Chang C, Du X, Hong M, Li X, Liu Q, Wang W, Xu N, Yang H, Lu B, Yin H, Wu L, Suo S, Zhao Q, Xiao Z, Jin J. Safety and efficacy of jaktinib (a novel JAK inhibitor) in patients with myelofibrosis who are intolerant to ruxolitinib: A single-arm, open-label, phase 2, multicenter study. Am J Hematol. 2023 Oct;98(10):1588-1597. doi: 10.1002/ajh.27033. Epub 2023 Jul 20. PMID 37470365
- [Background] Zhang Y, Zhou H, Suo S, Zhuang J, Yang L, He A, Liu Q, Du X, Gao S, Li Y, Li Y, Chen Y, Wu W, Zhu H, He G, Hong M, Jiang Q, Jiang Z, Jing H, Wang J, Xu N, Yue L, Zheng C, Zhou Z, Jin C, Li X, Liu L, Xu Y, Wu D, Zhang F, Zhang J, Wu L, Yin H, Lv B, Xiao Z, Jin J. Evaluation of gecacitinib vs hydroxyurea in patients with intermediate-2 or high-risk myelofibrosis: final analysis results from a randomized phase 3 study. Blood Cancer J. 2024 Dec 18;14(1):216. doi: 10.1038/s41408-024-01202-8. PMID 39695117
- [Background] Zhang Y, Zhang Q, Liu Q, Dang H, Gao S, Wang W, Zhou H, Chen Y, Ma L, Wang J, Yang H, Lu B, Yin H, Wu L, Suo S, Zhao Q, Tong H, Jin J. Safety and efficacy of jaktinib (a novel JAK inhibitor) in patients with myelofibrosis who are relapsed or refractory to ruxolitinib: A single-arm, open-label, phase 2, multicenter study. Am J Hematol. 2023 Oct;98(10):1579-1587. doi: 10.1002/ajh.27031. Epub 2023 Jul 19. PMID 37466271